CLINICAL TRIAL: NCT02873884
Title: Impact of Case-management on Therapeutic Alliance With First Episode Psychosis Patients (CAMAT)
Acronym: CAMAT
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: University Hospital, Caen (Other)
Responsible Party: Sponsor
Other Study IDs: CAMAT
Record Dates: First submitted 2016-08-17; First posted 2016-08-22 (Estimated); Last update posted 2019-04-22 (Actual); Status verified 2019-04

CONDITIONS: Psychotic Disorders
MeSH Terms: conditions — Psychotic Disorders | interventions — Case Management

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 6 Months

GROUPS / COHORTS (2):
- case-management: Patients will meet the case-manager 5 times per month during 1h30 in community living
  Interventions: Behavioral: Case-management
- traditional nursing: Patients will meet the case-manager 2 times per month during 1h00 in hospital

INTERVENTIONS:
Behavioral: Case-management
  Groups: case-management

SUMMARY:
The first aim of this study is to test the effect of the case management on the evolution of therapeutic alliance in patients with first episode psychosis in comparison with traditional nursing. The second aim is to test the effect of case management on nurses' well-being in comparison with traditional nursing. The third objective aims to show if therapeutic alliance is associated with insight in patients and with clinical and demographic data.

ELIGIBILITY:
Inclusion Criteria:

* Age between 16 and 30 years
* First episode psychosis diagnosis according to DSM-5 criteria

Exclusion Criteria:

* Lees of 16 years or more than 30 years
* Not fulfilling DSM-5 criteria for first episode psychosis
* Any treatment with the psychologist or the psychiatrist of the team

Ages: 16 Years to 30 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Study Population: First episode psychosis patients
Sampling Method: Probability Sample
Enrollment: 30 (Estimated)
Dates: Start 2016-11 (Actual); Primary Completion 2019-11 (Estimated); Study Completion 2019-11 (Estimated)

PRIMARY OUTCOMES:
Work alliance inventory | 6 months

SECONDARY OUTCOMES:
Birchwood insight scale | 6 months
Scale to assess Unawareness of Mental Disorder | 6 months
Well-being at work scale | 6 months

CONTACTS AND LOCATIONS:
Locations (1):
- CHU de Caen, Caen, France